CLINICAL TRIAL: NCT01007851
Title: Single Dose Gonadotropin-releasing Hormone (GnRH) Agonist Administration in the Luteal Phase of GnRH Antagonist Stimulated ICSI-ET Cycles
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lower than anticipated recruitment
Sponsor: V.K.V. American Hospital, Istanbul (Other)
Other Study IDs: AH-48/07
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2009-11-04 (Estimated); Status verified 2009-11

CONDITIONS: Infertility
Keywords: GnRH agonist; GnRH antagonist; IVF; ICSI; assisted reproduction; luteal phase
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate; Sodium Chloride

ARMS (2):
- GnRH agonist (Experimental)
  Interventions: Drug: triptorelin acetate
- Saline (Placebo Comparator)
  Interventions: Drug: NaCl %0.9

INTERVENTIONS:
Drug: triptorelin acetate — single dose of 0.1 mg triptorelin subcutaneous injection on the 3rd day after embryo transfer
  Arms: GnRH agonist
Drug: NaCl %0.9 — 0.1 ml sterile saline sc injection 3 days after embryo transfer
  Arms: Saline

SUMMARY:
GnRH agonist administration in the luteal phase was reported to beneficially affect clinical outcome of ICSI-ET cycles. This randomized controlled trial evaluates the effect of a single dose GnRH agonist administered in the luteal phase on the outcome of ICSI - ET cycles stimulated with the fixed GnRH antagonist protocol. Women undergoing embryo transfer following controlled ovarian hyperstimulation with a fixed GnRH antagonist protocol were included. In addition to routine luteal phase support with progesterone women were randomized to receive a single dose of GnRH agonist or placebo on the sixth day after ICSI.Ongoing pregnancy rate was the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing embryo transfer following controlled ovarian hyperstimulation with a fixed GnRH antagonist protocol, oocyte pick-up and ICSI.
* Embryo transfer performed on day 3

Exclusion Criteria:

* Participation in another trial that was being conducted in our unit at the same time.
* Preimplantation genetic screening cycles.
* Day 5 embryo transfers.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2006-09; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy beyond 20th gestational week

SECONDARY OUTCOMES:
clinical pregnancy rate
Embryo implantation rate

CONTACTS AND LOCATIONS:
Locations (1):
- American Hospital, Istanbul, Turkey (Türkiye)